CLINICAL TRIAL: NCT00458042
Title: Transitioning To Intravenous Remodulin® (Treprostinil Sodium) From Inhaled Iloprost (Ventavis®) in Patients With Pulmonary Arterial Hypertension: Safety, Efficacy and Treatment Satisfaction
Brief Title: Transitioning To IV Remodulin From Ventavis in Patients With PAH: Safety, Efficacy and Treatment Satisfaction
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low Enrollment
Sponsor: United Therapeutics (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIV-PH-412
Record Dates: First submitted 2007-04-05; First posted 2007-04-09 (Estimated); Last update posted 2007-11-12 (Estimated); Status verified 2007-11

CONDITIONS: Hypertension, Pulmonary
Keywords: Ventavis; iloporst; Remodulin; treprostinil; PAH; prostacyclin
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: treprostinil sodium

SUMMARY:
The purpose of this study is to compare the effects of switching from inhaled Ventavis to intravenous Remodulin in PAH patients who are considered to be failing inhaled Ventavis therapy. This study is intended to provide information on the safe transition from Ventavis to Remodulin as well as the impact intravenous Remodulin may have on overall quality of life and treatment satisfaction compared to Ventavis.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH), which is defined as an elevation in pulmonary arterial pressure and pulmonary vascular resistance, is a severe hemodynamic abnormality common to a variety of diseases and syndromes. Elevation in pulmonary arterial pressure causes an increase in right ventricular afterload, impairing right ventricular function and ultimately leading to inactivity and death. The goal of PAH treatment is to lengthen survival time, to ameliorate symptoms of PAH and to improve quality of life (QOL).

Remodulin (treprostinil sodium), a prostacyclin analog, possesses potent pulmonary and systemic vasodilatory and platelet anti-aggregatory actions in vitro and in vivo. Remodulin is an approved pharmacotherapy for PAH delivered as either a continuous subcutaneous infusion or intravenous infusion. Ventavis (iloprost)is an inhaled prostacyclin analogue with similar properties to Remodulin. In December 2004, Ventavis was approved for use in the United States by the FDA for the treatment of pulmonary arterial hypertension (WHO Group I) for patients with NYHA III or IV symptoms.

As the PAH community gains experience with the use of inhaled Ventavis, questions have arisen as to how to transition a patient on inhaled Ventavis to Remodulin in the presence of worsening symptoms or at a patient's request related to dissatisfaction with the frequency of daily treatments. This study will examine effects of switching from Ventavis to IV Remodulin and compare changes in exercise capacity, safety, HRQOL and treatment satisfactions.

Participation will last up to 12 weeks. Study procedures include routine blood tests, medical history, physical exams, disease evaluation, exercise tests and patient questionnaires. Participates will have 4 clinic visits during the study and will spend at least one night in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 years and 65 years of age
* WHO Class II-III
* Diagnosis of one of the following Group I WHO clinical classifications: Idiopathic or familial pulmonary arterial hypertension (PAH) or PAH associated with a collagen vascular disease or PAH associated with congenital systemic-to-pulmonary shunt repaired greater than 5 years prior to study entry or PAH associated with portal hypertension with mild or moderate hepatic dysfunction or PAH associated with drugs or toxins.
* Receiving inhaled iloprost for at least two months prior to screening or prior to treatment discontinuation.
* May have discontinued iloprost treatment against medical advice up to thirty days prior to screening
* Be mentally and physically capable of learning to administer Remodulin using an intravenous infusion pump.

Exclusion Criteria:

* Be a nursing or pregnant woman
* Have any PAH medication, other than inhaled iloprost, discontinued within the week prior to study entry.
* Received any prostacyclin or prostacyclin analog except iloprost in the past 3 months.
* Previous history of significant parenchymal lung disease
* Have any other type of PAH including but not limited to PAH related to thrombotic or embolic disease
* Have evidence of left-sided heart disease
* Musculoskeletal disorder (e.g. arthritis, artificial leg, etc.) or any other disease, which is thought to limit ambulation, or be connected to a machine, which is not portable.
* Uncontrolled systemic hypertension or chronic renal insufficiency
* Use of an investigational drug within the past 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2007-03; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Primary Outcomes: Change in distance traversed during the six minute walk test at 8 weeks;
Adverse events

SECONDARY OUTCOMES:
Secondary Outcomes: Borg dyspnea score immediately after the six minute walk test;
WHO functional classification;
Symptoms of PAH;
Specific prostacyclin side effects;
Total weekly time spent with specific activities associated with intravenous Remodulin therapy compared to the total weekly time spent on specific activities with inhaled Ventavis;
Score on treatment satisfaction scale;
Score on quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Hyong (Nick) Kim, MD, Principal Investigator — UCSD Medical Center
Locations (2):
- United States (2):
  - UCSD Medical Center Thornton Hospital, La Jolla, California
  - UCSD Medical Center Hillcrest Campus, San Diego, California